CLINICAL TRIAL: NCT05367310
Title: Effect of Breastfeeding on Lipid Profile and Cardiovascular Risk Markers in Women With Familial Hypercholesterolemia (FH-FEMINA)
Brief Title: Effect of Breastfeeding on Lipid Profile and Cardiovascular Risk Markers in Women With Familial Hypercholesterolemia
Acronym: FH-FEMINA
Status: Active, not recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Kirsten Bjørklund Holven, Professor, Oslo University Hospital
Other Study IDs: 395816
Record Dates: First submitted 2022-04-30; First posted 2022-05-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Familial Hypercholesterolemia
Keywords: Breastfeeding; Cardiovascular disease; Pregnancy; Lipid profile; Women
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Breast Feeding; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma, peripheral blood mononuclear cells, breastmilk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with familial hypercholesterolemia: Women with familial hypercholesterolemia
- Women without hypercholesterolemia: Women without hypercholesterolemia

SUMMARY:
The study aims to investigate the effects of breastfeeding on lipid profile and cardiovascular risk markers in women with familial hypercholesterolemia (FH) compared to women without FH. Women with FH will be recruited in Norway, the Netherlands, and the Czech Republic. Women without FH will be recruited in Norway.

Women with and without FH who are pregnant or planning pregnancy will be recruited, and will be invited to repeated study visits from the end of pregnancy and through the first year after delivery. Blood samples and data on anthropometry, health, pregnancy, lifestyle and diet will be collected. Statin transfer into breast milk will also be measured in breast milk samples collected when the women end breastfeeding the child and start statin treatment.

DETAILED DESCRIPTION:
Patients with familial hypercholesterolemia (FH) have elevated plasma levels of LDL-cholesterol from first years of life. Cholesterol burden through life defines risk of cardiovascular disease. In women with FH, cholesterol levels increase during pregnancy both due to physiological changes as well as discontinuation of cholesterol lowering medication during planning of pregnancy, during the pregnancy and during breastfeeding. Few studies on the effects of breastfeeding on lipid profile in women with FH exists. There is also limited data on whether and to what extent the cholesterol lowering statins transfer to breast milk.

The study aims to investigate the effects of breastfeeding on lipid profile and cardiovascular risk markers in women with familial hypercholesterolemia (FH) compared to women without FH.

Women with and without FH who are pregnant or planning pregnancy will be recruited, and will be invited to repeated study visits from the end of pregnancy and through the first year after delivery. Blood samples and data on anthropometry, health, pregnancy, lifestyle and diet will be collected. Statin transfer into breast milk will also be measured in breast milk samples collected when the FH women end breastfeeding the child and start statin treatment.

ELIGIBILITY:
Inclusion Criteria for women with FH:

1. age 18 years or older,
2. confirmed diagnosis of FH through genetic testing or clinical assessment based on the Dutch Lipid Clinic Network,
3. singleton pregnancy in the third trimester,
4. a sufficient command of Norwegian, Dutch, Czech or English language.

Exclusion Criteria for women with FH:

* Not filling the inclusion criteria.

Inclusion Criteria for women without FH:

1. age 18 years or older,
2. singleton pregnancy in the third trimester,
3. a sufficient command of Norwegian or English language.

Exclusion Criteria for women without FH:

1. known pre-pregnancy hypercholesterolemia,
2. a history of ASCVD.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with and without familial hypercholesterolemia (FH)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in serum lipid profile (total cholesterol, LDL-C, HDL-C, triglycerides, lipoprotein(a)) from 2-4 weeks postpartum up to 12 months postpartum (absolute and relative change). | Up to 12 months after delivery or end of breastfeeding period
  Investigate the change in lipid profile (total cholesterol, LDL-cholesterol, HDL-cholesterol and triglycerides) in women with and without familial hypercholesterolemia, by blood sampling at repeated time points during breastfeeding period.

SECONDARY OUTCOMES:
Association between breastfeeding (yes/no, exclusive/partial, frequency, and duration) and inflammatory markers (e.g. C-reactive protein (CRP). | Up to 12 months after delivery or end of breastfeeding period
  Investigate the association between breastfeeding (yes/no, exclusive/partial, frequency, and duration) and inflammatory markers (e.g. C-reactive protein) in women with and without familial hypercholesterolemia. Measurements will be performed in both plasma/serum and in peripheral blood mononuclear cells (PBMC) (gene expression levels).
Association between breastfeeding (yes/no, exclusive/partial, frequency, and duration) and metabolic markers (e.g. glucose). | Up to 12 months after delivery or end of breastfeeding period
  Investigate the association between breastfeeding (yes/no, exclusive/partial, frequency, and duration) and metabolic markers (e.g. glucose) in women with and without familial hypercholesterolemia. Measurements will be performed in both plasma/serum.
Association between breastfeeding (yes/no, exclusive/partial, frequency, and duration) and maternal weight. | Up to 12 months after delivery or end of breastfeeding period
  Investigate the association between breastfeeding (yes/no, exclusive/partial, frequency, and duration) and maternal weight in women with and without familial hypercholesterolemia.
Investigate the breast milk composition (lipids and metabolites) throughout the breastfeeding period. | Up to 12 months after delivery or end of breastfeeding period
  Perform lipid profiling (lipidomics) and metabolite profiling (metabolomics) and analyze contaminants in breast milk samples of women with FH and without FH. Breast milk samples will be collected at repeated time points through breast feeding period
Investigate the concentration of statins in the breast milk and dried blood spot of the offspring of women with FH after start of lipid-lowering medication. | Repeated milk sampling up to one week after start of ordinary statin treatment.
  Investigate the concentration of statin (HMG-CoA reductase inhibitors) (e.g. atorvastatin, rosuvastatin) in breast milk and dried blood spot of the offspring, if possible when the women re-start ordinary treatment. Fewer samples are expected from this time point, as it may be challenging to synchronize the initiation of lipid-lowering treatment with the end of breastfeeding.
Investigate the concentration of total cholesterol and metabolic markers in dried blood spots collected at 12 months postpartum in offspring of women with FH | Measurement at infant age 12 months
  Investigate the concentration of total cholesterol and other metabolic markers in infants of women with FH, at 12 months of age, using dried blood spots (DBS).

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Holven, PhD, Principal Investigator — Oslo University Hospital
Locations (4):
- Czechia (2):
  - Centre of Cardiovascular Surgery and Transplantation, Brno
  - Third Department of Internal Medicine, General University Hospital, First Faculty of Medicine, Charles University, Prague
- Department of Internal Medicine, Erasmus MC Cardiovascular Institute, Rotterdam, Netherlands
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Klevmoen M, Mulder JWCM, Bogsrud MP, Retterstol K, Vesterbekkmo EK, Pedersen EKR, Freiberger T, Vrablik M, Vaclova M, Hovland A, Vethe NT, Brekke HK, Iversen PO, Veierod M, Roeters van Lennep J, Holven KB. Prospective study on breastfeeding, lipid profile and cardiovascular risk markers in women with familial hypercholesterolaemia: study protocol for the FH-FEMINA study. BMJ Open. 2025 Apr 27;15(4):e092208. doi: 10.1136/bmjopen-2024-092208. PMID 40288796